CLINICAL TRIAL: NCT04771676
Title: A Phase II Study of Intraperitoneal Injection of Oncolytic Viruses H101 for Patients With Refractory Malignant Ascites
Brief Title: Intraperitoneal Injection of Oncolytic Viruses H101 for Patients With Refractory Malignant Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012229-11
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Refractory Malignant Ascites

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncorine (H101) (Experimental): H101 diluted in 5ml 0.9% sodium chloride solution will be intraperitoneally injected through the drainage catheter. Each patient will receive a dose of 1.5×10^12 vp by i.p. administration on day 1 and 3.
  Interventions: Drug: Oncorine (H101)

INTERVENTIONS:
Drug: Oncorine (H101) — A modified human recombinant type 5 adenovirus with genetic modifications.

SUMMARY:
Assessment of effectiveness, safety and local immune activation of Oncolytic Viruses H101 in patients with refractory malignant ascites.

DETAILED DESCRIPTION:
This study is to evaluate the effectiveness of local immune activation, and safety in patients with refractory malignant ascites after Intraperitoneal injection of oncolytic Viruses H101.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Histologically diagnosed solid tumor malignancy.
* Malignant peritoneal ascites confirmed by cytologic examination.
* Failures from chemotherapy or other anti-cancer therapy or standard chemotherapy was no longer feasible.
* Cooperative Oncology Group-Status (ECOG Status) ≤ 2.
* life expectancy >8 weeks
* Estimated ascites volume >1 L by CT scan.
* At least one symptomatic paracentesis within 4 weeks as well as an objectively verified, clinical need for a second paracentesis
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/uL, platelets ≥60 x103u/L; Total bilirubin ≤ 3 x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula).
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* History or evidence of active autoimmune disease that requires systemic treatment.
* Acute or chronic active Hepatitis B or C infection or HIV infection.
* Previous (<4 weeks) or concurrent treatment with systemic or intraperitoneal chemotherapy or biological agents such as monoclonal antibodies.
* Concurrent severe illness such as active infection.
* Enteral feeding at study entry.
* Ileus within the previous 30 days
* >70% tumor infiltration of the liver or portal vein obstruction.
* Arterial or venous thromboembolic disease.
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results, including but not limited to:

  1. Known acute or chronic pancreatitis
  2. Active tuberculosis
  3. Any other active infection (viral, fungal or bacterial) requiring systemic therapy
  4. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
  5. History or clinical evidence of Central Nervous System (CNS) metastases. Exceptions for subjects who have completed local therapy. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS.
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year).[Acceptable methods of contraception are implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year).[Acceptable methods of contraception are implants, injectable contraceptives, combine d oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Time to repeat paracentesis (TTRP) | max 6 months
  Defined as the number of days between the first paracentesis (baseline) and the subsequent repeat paracentesis.

SECONDARY OUTCOMES:
Analysis of adverse events | max 6 months
  Toxicity were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
  All serious and non-serious adverse events that occur after enrollment through 30 (+7) days after the last administration of H101 will be recorded
Paracentesis free survival (PaFS) | max 6 months
  Difined as the time from the date of first paracentesis to the repeat paracentesis or death.
60-day frequency of paracentesis | max 6 months
  Defined as frequency of paracentesis during the first 60 days.
Overall survival (OS) | max 6 months
  Defined as the time from the date of patient enrollment until the date of death from any cause.
Change from baseline local and systemic immune effects after H101 intraperitoneal injections | at baseline, 3-, 7, 14 days after injection
  Detection of immune activation in malignant ascites and blood will be assessed by single cell sequencing and Mass Cytometry (CyTOF).

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China